CLINICAL TRIAL: NCT01917240
Title: Evaluation of the Impact of Monophasic vs. Sequential Media on the Reproductive Potential of Embryos Undergoing in Vitro Fertilization (IVF)
Brief Title: Sequential vs. Monophasic Media Impact Trial (SuMMIT)
Acronym: SuMMIT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RMA-2013-02
Record Dates: First submitted 2013-07-18; First posted 2013-08-06 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Infertility
Keywords: Monophasic; Sequential; Media
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Monophasic Media (Experimental): Half of each patient's embryos will be randomly assigned to grow in monophasic media & the other half in sequential media. All embryos will undergo CCS & the best euploid embryo from each group will be transferred (DET). If there are only euploid embryos from one group, pt will have SET only (fresh or frozen)
  Interventions: Other: Comprehensive Chromosome Screening
- Sequential Media (Placebo Comparator): Half of each patient's embryos will be randomly assigned to grow in monophasic media & the other half in sequential media. All embryos will undergo CCS & the best euploid embryo from each group will be transferred (DET). If there are only euploid embryos from one group, pt will have SET only (fresh or frozen)
  Interventions: Other: Comprehensive Chromosome Screening

INTERVENTIONS:
Other: Comprehensive Chromosome Screening — On day 5 or 6 of embryo development, all embryos will undergo a trophectoderm biopsy using the standardized technique, as according to standard laboratory protocol and without regard to study. Comprehensive Chromosome Screening (CCS) results will be available by the morning of day 6 if embryos are suitable for a fresh transfer which is the routine in our program.

SUMMARY:
To evaluate the impact of two FDA approved culture media on potential of human embryos resulting from IVF (sequential & monophasic media). Half of each patient's embryos will be randomly assigned to grow in monophasic media & the other half in sequential media. All embryos will undergo Comprehensive Chromosome Screening (CCS) & the best euploid embryo from each group will be transferred resulting in a double embryo transfer (DET). If there are only euploid embryos from one group, patient will have single embryo transfer (SET)(fresh or frozen).

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing IVF/CCS (no PGD banking)
* Patient meets ASRM guidelines for Double Embryo Transfer (DET)
* Donor Sperm OK
* AMH ≥ 1.2
* FSH ≤ 12
* BAFC ≥12
* Max 1 prior failed IVF cycle for patients 35-45 years old
* Patient <35 years old MUST have 1 prior failed IVF cycle

Exclusion Criteria:

* Chronic endometrial insufficiency
* Use of oocyte donor or gestational carriers
* Medical contraindications to Double Embryo Transfer (DET)
* Male Factor (<100,000 sperm or surgical sperm)
* Communicating hydrosalpinx (on HSG)
* Single gene disorders or sex selection

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2013-07; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Impact of monophasic vs. sequential media on the embryos produced from IVF on pregnancy rates | 2 years
  To assess if pregnancy rates are impacted by the type of culture media embryos produced by IVF are cultured in

CONTACTS AND LOCATIONS:
Overall Officials: Richard T. Scott, M.D., HCLD, Principal Investigator — Reproductive Medicine Associates of New Jersey
Locations (1):
- Reproductive Medicine Associates of New Jersey, Basking Ridge, New Jersey, United States

REFERENCES:
- [Derived] Werner MD, Hong KH, Franasiak JM, Forman EJ, Reda CV, Molinaro TA, Upham KM, Scott RT Jr. Sequential versus Monophasic Media Impact Trial (SuMMIT): a paired randomized controlled trial comparing a sequential media system to a monophasic medium. Fertil Steril. 2016 May;105(5):1215-1221. doi: 10.1016/j.fertnstert.2016.01.005. Epub 2016 Jan 27. PMID 26826274